CLINICAL TRIAL: NCT05342987
Title: The Relationship Between Delirium and Circadian Rhythm in Intensive Care Unit
Brief Title: Circadian Rhythm and Delirium in ICU
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021ZSYQ17
Record Dates: First submitted 2022-03-11; First posted 2022-04-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2022-03

CONDITIONS: Circadian Rhythm; Sleep Quality; Intensive Care Unit Delirium
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample will be taken to measure melatonin level using ELISA kit (produced by abcam)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims to investigate the status of circadian rhythm and sleep quality in ICU patients and their influence factors. And explore the pathway of circadian rhythm on ICU delirium.

The hypothesis of study is that icu patients experience circadian and sleep rhythm disorder, especially in patient who have delirium.

DETAILED DESCRIPTION:
Delirium is an acute and fluctuating alteration of mental state characterized by a disturbance in attention, level of consciousness and cognition. At present, there is no unified conclusion on the pathogenesis of delirium. There are many different hypotheses, such as the neuroinflammation hypothesis, the neuronal aging hypothesis, the oxidative stress hypothesis, the neurotransmitter hypothesis, the neuroendocrine hypothesis and the circadian rhythm disturbance hypothesis. Among them, the circadian rhythm disturbance hypothesis believes that the circadian rhythm disorder caused by various reasons, which leads to sleep disturbance and melatonin secretion disorder promotes the occurrence of acute cognitive impairment, which in turn leads to the occurrence of delirium. Circadian rhythm refers to the rhythm of any biological process in the human body that repeats and maintains within 24 hours without external stimulation. By far, the most common way to measure circadian rhythm is through vital signs rhythms, hormone secretion (cortisol and melatonin levels), and sleep-wake cycle.

Due to the special environment and treatment needs in ICU make patients' circadian rhythm easily broken, and produced a large latent harm to patients. Most studies are in the process of delirium and sleep research, selecting a small subgroup to evaluate the circadian rhythm indicators of patients, and the overall relationship between delirium and circadian rhythm is not clear.

Thus, the study aims to investigate the status of circadian rhythm and sleep quality in ICU patients and their influence factors, and explore the pathway of circadian rhythm action on ICU delirium.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18
* RASS>-4

Exclusion Criteria:

* History of mental or psychological illness
* The patient remained in coma or deep sedation
* Delirium was occurring at the time of admission
* Unable to fully participate in delirium testing, including blind, deaf, illiterate or inability to understand Chinese
* Neurosurgery and maternal patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 who are admitted to ICU will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes of melatonin level | Three time a day in 3, 8 and 16 clock on day 1 to day 3 and day 7 after admission in ICU
  Test Serum melatonin level
Sleep Quality | up to 14 days after admission in ICU
  Investigators screen sleep quality by Richards-Campbell Sleep Questionnaire
Changes of cortisol level | Three time a day in 0, 8 and 16 clock on day 1 to day 3 and day 7 after admission in ICU
  Test Serum cortisol level

SECONDARY OUTCOMES:
ICU delirium | up to 14 days after admission in ICU
  Investigators screen delirium by CAM-ICU twice a day, each time during day and night
patient outcome | up to 14 days after admission in ICU
  Mortality in ICU
LOS | up to 14 days after admission in ICU
  length of ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li J, Cai S, Liu X, Mei J, Pan W, Zhong M, Zhang Y. Circadian rhythm disturbance and delirium in ICU patients: a prospective cohort study. BMC Anesthesiol. 2023 Jun 13;23(1):203. doi: 10.1186/s12871-023-02163-4. PMID 37312021